CLINICAL TRIAL: NCT02683655
Title: Study of Apatinib in Metastatic Esophageal Cancer：A Open Label, Randomized Clinical Trial
Brief Title: Study of Apatinib in Metastatic Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huai'an First People's Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-E301
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apatinib 500mg qd p.o. (Experimental): Apatinib Mesylate Tablets 500 mg qd p.o. after the failure of chemotherapy or radiotherapy
  Interventions: Drug: Apatinib
- Apatinib 750mg qd p.o. (Experimental): Apatinib Mesylate Tablets 750 mg qd p.o. after the failure of chemotherapy or radiotherapy
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg qd p.o.
  Arms: Apatinib 500mg qd p.o.
Drug: Apatinib — Apatinib 750mg qd p.o.
  Arms: Apatinib 750mg qd p.o.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of apatinib in Metastatic Esophageal Cancer.

DETAILED DESCRIPTION:
Eligible patients will receive apatinib treatment until disease progression or intolerable toxicity or patients withdrawal of consent after the failure of chemotherapy or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to75 years old;
2. Pathologically diagnosed with metastatic esophageal squamous cell cancer with measurable metastases outside the stomach (measuring ≥ 10mm on spiral CT scan, satisfying the criteria in RECIST 1.1);
3. Failed in first-line chemotherapy or radiotherapy treatment;
4. ECOG PS of 0-1;
5. An expected survival of ≥ 3 months;
6. No treated by molecularly targeted therapy. If have received chemotherapy, radiotherapy or surgery, must ≥4 weeks, and adverse reactions or wound has been completely restored;
7. Major organ function has to meet the following criteria:

   ANC ≥ 1.5 × 109 / L; HB ≥ 90g / L; PLT ≥ 100 × 109 / L; ALB≥30g / L; TBIL≤1.5 times the upper limit of normal (ULN); ALT and AST<2 × ULN; Plasma Cr<1.5 × ULN
8. Patient has to voluntarily join the study and sign the Informed Consent Form for the study;
9. Researchers believe that patients can benefit;

Exclusion Criteria:

1. Pts with other malignant tumor at the same time or in the past.
2. Pregnant or lactating women;
3. Subjects with poor-controlled arterial hypertension (systolic blood pressure>150 mmHg and diastolic blood pressure>100 mm Hg) despite standard medical management; Coronary heart disease greater than ClassII; Echocardiography: LVEF (LVEF)<50%;
4. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
5. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 6 months;
6. Associated with CNS (central nervous system) metastases;
7. Abnormal Coagulation, with tendency of bleed;
8. With psychotropic drug abuse history and can't get rid of or mental disorder patients;
9. Anastomotic recurrence;
10. Participated in other clinical trials within 4 weeks;
11. Any other condition that might place the patient at undue risk or preclude a patient from completing the study;
12. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | An expected average of 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Huaian First People's Hospital, Huaian, Jiangsu, China